CLINICAL TRIAL: NCT06006910
Title: An Electronic Medical Record-Based Nudge Intervention to Reduce Low-Value Axillary Surgery in Older Women With ER+ Breast Cancer
Brief Title: Electronic Medical Record-Based Nudge to Reduce SLNB
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Priscilla McAuliffe, Assistant Professor, University of Pittsburgh Medical Center
Organization: University of Pittsburgh (Other)
Other Study IDs: 4040
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Estrogen-receptor-positive Breast Cancer
Keywords: Sentinel lymph node biopsy; Axillary surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Nudge Deployment into EHR: Rates of SLNB will be recorded for the 12 month period prior to nudge deployment.
  Interventions: Behavioral: No column-based nudge in the EHR
- Post-Nudge Deployment into EHR: Rates of SLNB will be recorded for the 12 month period following nudge deployment into the EHR.
  Interventions: Behavioral: Column-based nudge in the EHR

INTERVENTIONS:
Behavioral: Column-based nudge in the EHR — The nudge is a column in EPIC that flags patients coming to the clinic as a new visit with documented ER+ breast cancer. The nudge flag can pop up when hovered over to remind surgeons of the Choosing Wisely criteria and to consider omission of SLNB.
  Groups: Post-Nudge Deployment into EHR
Behavioral: No column-based nudge in the EHR — No intervention control period prior to nudge deployment.
  Groups: Pre-Nudge Deployment into EHR

SUMMARY:
The goal of this prospective, historically-controlled, quality improvement project is to determine whether and to what extent an electronic health record (EHR)-based nudge affects rates of sentinel lymph node biopsy (SLNB) in older women with ER+, early-stage, clinically node negative breast cancer.

DETAILED DESCRIPTION:
Society of Surgical Oncology (SSO) adopted a series of Choosing Wisely recommendations in an effort to reduce low-value surgeries. One such recommendation, first released in 2016, advocates against routine use of sentinel lymph node biopsy (SLNB) for axillary staging in older women (≥ 70 years old) with early-stage, estrogen receptor positive (ER+), clinically node-negative breast cancer. Data supporting this recommendation were largely retrospective in nature as there were no direct randomized trials testing de-escalation of SLNB in this population of patients. This has led to variability in de-implementation of SLNB, with rates of SLNB use still reaching 50%-60% in some centers.

To address this, the investigators designed an electronic medical record-based column nudge that flags patients meeting Choosing Wisely criteria for omission of SLNB. This was designed to target surgeons in the moments leading up to the first clinic visit with patients where surgical decision-making is planned. In this study, the investigators deployed the column nudge for a 12 month period.

The enrollment number reflects the number of surgeons participating in the study (whom the nudge was deployed to); it is anticipated this group of surgeons will see over 400 patients between the pre-nudge and post-nudge periods.

ELIGIBILITY:
Inclusion Criteria:

* early-stage (stages I-III) breast cancer
* clinically node-negative
* ER+ and/or PR+, HER2 not-amplified
* non-metastatic at diagnosis

Exclusion Criteria:

* under 70 years of age
* breast cancer is that is not ER+ or PR+

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Women 70 years or older with ER+/PR+ and HER2-, early-stage, clinically node negative breast cancer
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Rate of SLNB after nudge deployment into the EHR | 12 months
  We will record the rate of SLNB use (yes/no for if the surgeon performed the surgery) per month over a 12 month intervention period. Rate of SLNB after nudge deployment will be compared to rate of SLNB before nudge deployment.

SECONDARY OUTCOMES:
Acceptability of Intervention (AIM) [Survey] | 2 weeks prior to nudge deployment into the EHR
  AIM is a validated, 4-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.
Intervention Appropriateness Measure (IAM) [Survey] | 2 weeks prior to nudge deployment into the EHR
  AIM is a validated, 4-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.
Feasibility of Intervention Measure (FIM) [Survey] | 2 weeks prior to nudge deployment into the EHR
  AIM is a validated, 4-item survey with all items measured on a 5-point Likert scale (Completely Disagree [1] - Completely Agree [5]), scored as a mean. The median score across all participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla F McAuliffe, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carleton N, Oesterreich S, Marroquin OC, Diego EJ, Tseng GC, Lee AV, McAuliffe PF. Is the Choosing Wisely Recommendation for Omission of Sentinel Lymph Node Biopsy Applicable for Invasive Lobular Carcinoma? Ann Surg Oncol. 2022 Sep;29(9):5379-5382. doi: 10.1245/s10434-022-12003-3. Epub 2022 Jun 13. No abstract available. PMID 35697956
- [Background] Carleton N, Zou J, Fang Y, Koscumb SE, Shah OS, Chen F, Beriwal S, Diego EJ, Brufsky AM, Oesterreich S, Shapiro SD, Ferris R, Emens LA, Tseng G, Marroquin OC, Lee AV, McAuliffe PF. Outcomes After Sentinel Lymph Node Biopsy and Radiotherapy in Older Women With Early-Stage, Estrogen Receptor-Positive Breast Cancer. JAMA Netw Open. 2021 Apr 1;4(4):e216322. doi: 10.1001/jamanetworkopen.2021.6322. PMID 33856473
- [Derived] Carleton N, Radomski TR, Li D, Zou J, Harris J, Hamm M, Wang Z, Saadawi G, Fischer GS, Arnold J, Cowher MS, Lupinacci K, Sabih Q, Steiman J, Johnson RR, Soran A, Diego EJ, Oesterreich S, Tseng G, Lee AV, McAuliffe PF. Electronic Health Record-Based Nudge Intervention and Axillary Surgery in Older Women With Breast Cancer: A Nonrandomized Controlled Trial. JAMA Surg. 2024 Oct 1;159(10):1117-1125. doi: 10.1001/jamasurg.2024.2407. PMID 39018053